CLINICAL TRIAL: NCT06218212
Title: The Effect of Renastart Formula Supplementation on Serum Electrolytes in Children With Acute Kidney Injury
Brief Title: The Effect of Renastart Formula Supplementation in Children With Acute Kidney Injury in Maintaining Normal Serum Electrolytes Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, lecturer of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 643/ 2021
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Calcium Carbonate; polystyrene sulfonic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 patients with AKI and acute on top of CKD who will be treated by electrolytes binders. (Active Comparator): they will start calcium carbonate (phosphorus binder) with dosage 45-65 mg/kg/day orally with / or sodium polystyrene sulfonate (potassium binder) with dosage 0.5-1mg/kg/day orally.
  Interventions: Drug: calcium carbonate (phosphorus binder) with / or sodium polystyrene sulfonate (potassium binder) with dosage 0.5-1mg/kg/day orally.
- Arm 2 patients with AKI and acute on top of CKD who will be treated by Renastart formula. (Experimental): * Renastart formula will be used with breast milk, standard infant formula or with diet.
  * Preparation: Adding one level scoop of Renastart to 30 ml water.
  * Renastart formula will be started to represent ¼ recommended daily allowance of daily caloric intake and the dose will be adjusted according to serum electrolyte levels.
  Interventions: Dietary Supplement: Renastart formula

INTERVENTIONS:
Dietary Supplement: Renastart formula — * Renastart formula is an artificial formula is made by Vitaflo USA, Nestle Health Science Company.
  * Renastart formula preparation: Adding one level scoop of Renastart to 30 ml water.
  * Renastart formula will be used with breast milk, standard infant formula, standard pediatric infant feed and/ or mixed with diet.
  * Renastart formula dosage will be adjusted to be 1/4 Renastart and 3/4 breast milk, standard infant formula or standard pediatric infant daily caloric feed ratio.
  * Readjusting dosage ratio according to serum electrolytes levels especially potassium.
  Arms: Arm 2 patients with AKI and acute on top of CKD who will be treated by Renastart formula.
Drug: calcium carbonate (phosphorus binder) with / or sodium polystyrene sulfonate (potassium binder) with dosage 0.5-1mg/kg/day orally. — calcium carbonate (phosphorus binder) in dosage of 45-65 mg/kg/day orally with / or sodium polystyrene sulfonate (potassium binder) in dosage of 0.5-1mg/kg/day orally.
  Arms: Arm 1 patients with AKI and acute on top of CKD who will be treated by electrolytes binders.

SUMMARY:
This clinical trial will evaluate Renastart formula effectiveness in children with acute kidney injury (AKI) and acute on top of chronic kidney disease (CKD), in maintaining normal serum electrolytes levels without using electrolyte binders,24 patients will be recruited from Pediatric Nephrology Unit (PNU), Children's Hospital, Ain Shams University, they will be assigned randomly in to two arms, arm 1 including patients who will be treated by electrolytes binders, arm 2 including patients who will be treated by Renastart formula, after initial assessment serum electrolyte evaluation will be followed up monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

•Infants and Children with AKI and acute on top of CKD Suffering from hyperkalemia and/or hyperphosphatemia at Pediatric Nephrology Unit (PNU), Children's Hospital, Ain Shams University Hospitals.

Exclusion Criteria:

* Patients are on dialysis.
* Pediatric patients with coexisting another medical problems and different risk factors which can affect serum electrolytes such as: Constipation, high volume blood transfusion and Diabetes medications disrupt potassium balance e.g., ACEI, ARBS and Diuretics.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness and tolerability of Renastart formula in children with AKI and acute on top of CKD to correct and maintain normal serum levels of electrolytes. | monthly for 3 months
  serum electrolytes

CONTACTS AND LOCATIONS:
Overall Officials: Haya E Ibrahim, MD, Principal Investigator — lecturer of pediatrics,Faculty of Medicine, Ain shams University
Locations (1):
- Faculty of Medicine-Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided